CLINICAL TRIAL: NCT06483698
Title: Real-world Clinical Outcomes of Patients With Early-stage Lung Cancer After the Surgery: A Retrospective Multi-center Study (EarlyLC-RW)
Brief Title: Real-world Clinical Outcomes of Patients With Early-stage Lung Cancer After the Surgery
Acronym: EarlyLC-RW
Status: Recruiting | Type: Observational
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 23/516-4259
Record Dates: First submitted 2024-03-12; First posted 2024-07-03 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-04

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Anterior Temporal Lobectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sublobar resection group: Patients in this group have received Sublobar resection.
  Interventions: Other: Sublobar resection
- Lobectomy group: Patients in this group have received lobectomy.
  Interventions: Other: Lobectomy

INTERVENTIONS:
Other: Sublobar resection — Sublobar resection is a series of surgical approaches for lung cancer.
  Groups: Sublobar resection group
Other: Lobectomy — Lobectomy is the surgical approach for lung cancer.
  Groups: Lobectomy group

SUMMARY:
The goal of this observational study is to evaluate the efficacy and long-term clinical outcomes of early-stage lung cancer patients who have received surgery using the real-world data. The main questions it aims to answer are:

* What is the best surgical strategy for patients with early-stage lung cancer?
* What are the risk factors for early-stage lung cancer? Participants will receive surgery and the study will analyze the real-world data.

DETAILED DESCRIPTION:
This observational study aims to comprehensively evaluate the effectiveness and long-term clinical outcomes of surgical interventions in early-stage lung cancer patients, utilizing real-world data.

Central to this investigation are two key questions:

* What is the optimal surgical approach for managing early-stage lung cancer?
* What are the primary risk factors associated with the development of early-stage lung cancer? Participants will undergo surgical procedures, and through rigorous analysis of real-world data, this study endeavors to provide nuanced insights into these fundamental queries, fostering advancements in clinical decision-making and patient management strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 85;
2. Did not receive neoadjuvant therapy before surgery;
3. No history of radiation therapy;
4. Eastern Cooperative Oncology Group (ECOG) score is 0-1;
5. Have complete clinically relevant information including imaging data;
6. All patients underwent relevant preoperative examinations;
7. Stage I lung cancer (International Association for the Study of Lung Cancer/The Union for International Cancer Control staging eighth edition);

Exclusion Criteria:

1. Have previously received chemotherapy, radiotherapy and other anti-tumor therapy;
2. Data loss and error in medical records due to human/objective reasons.

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with lung cancer who have received surgery.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2034-12 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival(DFS) | Defined as the time from the date of surgery until the date of first documented progression or death (by any cause in the absence of recurrence), whichever came first, assessed up to 10 years.
  Defined as the time from the date of randomization until the date of disease recurrence or death (by any cause in the absence of recurrence).

SECONDARY OUTCOMES:
Overall Survival (OS) | From date of diagnosis until the date of death from any cause, whichever came first, assessed up to 10 years.
  OS is defined as the time from surgery time until death from any cause.
5-year Overall Survival (overall survival) Rate | From date of surgery until date of death due to any cause. Assessed at 5 years.
  The time from surgery time until death from any cause, estimated from a Kaplan Meier plot of OS at the time of the primary analysis.
Patterns of Relapse | Within 10 years after surgery
  Relapse was defined as disease recurrence at any site.
Perioperative Complication rate | Within 6 months after surgery
  Complications after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Shugeng Gao, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Shugeng Gao, Beijing, Beijing Municipality, China